CLINICAL TRIAL: NCT05636501
Title: Dose Reduction and Discontinuation of Prednisolone Using Structured Treat-to-target Taper in Patients With Polymyalgia Rheumatica
Brief Title: Treat-to-target Prednisolon Taper in Patients With Polymyalgia Rheumatica
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Horsens Hospital (Other); Regionshospitalet Silkeborg (Other); Gødstrup Hospital (Other); Regionshospital Nordjylland (Other Government); Aalborg University Hospital (Other); Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Kresten Krarup Keller, MD associate professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T2T PMR
Record Dates: First submitted 2022-11-10; First posted 2022-12-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treat-to-target Prednisolone Taper (Active Comparator): Patients randomized to the "Treat-to-target" group is prescribed with a systematic prednisolone taper according to a specific scheme. The starting dose can be increased if remission is not reached initially or in case of relapse, folloved by taper according to the specific scheme. A nurse will make a minimum of 5 phone consultations the first year, and hereafter minimum every 3 months.
  Interventions: Other: Treat-to-target Prednisolone Taper
- Usual Care (Placebo Comparator): Patients randomized to "usual care" are dismissed from the hospital after the diagnosis and the prednisolone taper are subsequently performed by discretion of the patient's general practitioner.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Treat-to-target Prednisolone Taper — Systematic prednisolone taper
  Arms: Treat-to-target Prednisolone Taper
Other: Usual care — Prednisolone taper performed by discretion of the patient's general practitioner.
  Arms: Usual Care

SUMMARY:
Polymyalgia rheumatica (PMR) has an incidence of approximately 1000/10^6 for persons more than 50 years. Treatment with prednisolone carries several significant adverse effects, and it is therefore essential to taper prednisolone as fast as possible. Systematic treatment strategies (treat-to-target) is the most important improvement of disease management for other rheumatic diseases such as rheumatoid arthritis in the last decades. Thus, the purpose is to investigate benefits and harms associated with a nurce led systematic prednisolone taper strategy at the department of rheumatology compared to individual treatment by discretion of the general practitioner. It is a 1-year open label randomised trial with a 1-year extension in 120 treatment naïve patients with PMR.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with PMR according to the EULAR criteria for PMR.
* No sign of GCA on ultrasonography of the temporal and axillary arteries.
* Age over 50 years.
* Danish spoken and written language skills sufficient to fill out questionnaires.

Exclusion Criteria:

* Peroral, intraarticular or intramuscular application of glucocorticoids within the last month.
* Previous prednisolone treatment for GCA/PMR.
* Unable to give consent.
* Symptoms of GCA (newly onset-headache, tenderness of the temporal artery, jaw claudication, vision disturbances).
* Active malignant cancers within the last 5 years (except basal cell carcinoma).
* Other inflammatory rheumatic diseases (eg. rheumatoid arthritis, polymyositis, spondyloarthritis, psoriatic arthritits, gout).
* Uncontrolled diseases (eg severe active asthma, cardiac disease with NYHA class IV)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in prednisolone free remission 52 weeks from baseline | 52 weeks
  Proportion of patients in prednisolone free remission 52 weeks from baseline

SECONDARY OUTCOMES:
Change in prednisolone dose from baseline to week 52 | 52 weeks
  Change in prednisolone dose from baseline to week 52. Key secondary.
Proportion of GCA patients diagnosed during the first 52 weeks | 52 weeks
  Proportion of GCA patients diagnosed during the first 52 weeks. Key secondary
Self-reported number of relapses during the first 52 weeks | 52 weeks
  Self-reported number of relapses during the first 52 weeks (assessed by increase in symptoms and an increase in prednisolone dosage). Key secondary
Change in patient-reported global visual analogue scale (VAS) from baseline to week 52 | 52 weeks
  Change in patient-reported global VAS from baseline to week 52. Scale 0-10, 10 is worse. Key secondary
Change in polymyalgia rheumatica activity score (PMR-AS) from baseline to week 52 | 52 weeks
  Change in PMR-AS from baseline to week 52. scale 0-indefinitely. High score is worse. Secondary
Proportion of patients with an undiagnosed vasculitis assessed by ultrasound at week 52 Proportion of patients with an undiagnosed vasculitis assessed by ultrasound at week 52 | 52 weeks
  Proportion of patients with an undiagnosed vasculitis assessed by ultrasound at week 52. Secondary
Changes in short form (SF)-36 mental component summary (MCS) from baseline to week 52 | 52 weeks
  Changes in SF-36 MCS from baseline to week 52. Secondary
Changes in short form (SF)-36 physical component summary (PCS) from baseline to week 52 | 52 weeks
  Changes in SF-36 PCS from baseline to week 52. Secondary
Changes in health assessment questionnaire disability index (HAQ-DI) from baseline to week 52 | 52 weeks
  Changes in HAQ-DI from baseline to week 52. High score is worse. Secondary
Changes in patient reported polymyalgia rheumatica visual analog scale (PMR VAS) from baseline to week 52 | 52 weeks
  Changes in patient reported PMR VAS from baseline to week 52. High score is worse. Secondary
Changes in patient reported fatigue visal analog scale (VAS) from baseline to week 52 | 52 weeks
  Changes in patient reported fatigue VAS from baseline to week 52. Higher is worse. Secondary
Changes in patient reported stiffness visual analog scale (VAS) from baseline to week 52 | 52 weeks
  Changes in patient reported stiffness VAS from baseline to week 52. Higher is worse. Secondary
Changes in patient reported duration of morning stiffness from baseline to week 52 | 52 weeks
  Changes in patient reported duration of morning stiffness from baseline to week 52. Secondary
Proportion of patients where baseline DXA scan are performed during the first 3 months after baseline visit | 3 months
  Proportion of patients where baseline DXA scan are performed during the first 3 months after baseline visit. Secondary
Proportion of patients where HgbA1C blood samples are taken during the first 52 weeks | 52 weeks
  Proportion of patients where HgbA1C blood samples are taken during the first 52 weeks. Secondary
Frequency of patient reported adverse effects and comorbidities related to prednisolone treatment after 13, 26, 39 and 52 weeks | 52 weeks
  Frequency of patient reported adverse effects and comorbidities related to prednisolone treatment after 13, 26, 39 and 52 weeks. Secondary.
Proportion of patients with patient reported infections during the first 52 weeks | 52 weeks
  Proportion of patients with patient reported infections during the first 52 weeks. Secondary.

CONTACTS AND LOCATIONS:
Overall Officials: Kresten Keller, Principal Investigator — Aarhus University Hospital
Locations (6):
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Department of Rheumatology, Aarhus
  - Gødstrup Regional Hospital, Herning
  - Hjørring Regional Hospital, Hjørring
  - Horsens Regional Hospital, Horsens
  - Silkeborg Regional Hospital, Silkeborg

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in the publications
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication, and 2 years.
Access Criteria: By resonably request.

DOCUMENTS (2):
  • Study Protocol (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT05636501/Prot_001.pdf
  • Statistical Analysis Plan (2025-06-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT05636501/SAP_000.pdf